CLINICAL TRIAL: NCT02829372
Title: A Phase 1, First-in-man, Multicenter, Open-label, Dose-escalation Study of Single-agent GBR 1302 in Subjects With HER2 Positive Cancers
Brief Title: Phase 1 Study of Single Agent GBR 1302 in Subjects With HER2 Positive Cancers
Acronym: GBR 1302-101
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention
Sponsor: Ichnos Sciences SA (Industry)
Collaborators: Glenmark Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBR 1302-101; 2015-002926-38 (EudraCT Number)
Record Dates: First submitted 2016-07-01; First posted 2016-07-12 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: HER2 Expressing Solid Tumours

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GBR 1302 (Experimental): Dose escalation
  Interventions: Drug: CD3/HER2 bispecific monoclonal antibody

INTERVENTIONS:
Drug: CD3/HER2 bispecific monoclonal antibody — Increasing doses, IV on day 1 and 15 of each 28 day cycle

SUMMARY:
The purpose of this study is to determine the safety profile and maximum tolerable dose (MTD) of GBR 1302 monotherapy in subjects with HER2 positive cancers

ELIGIBILITY:
Inclusion Criteria:

1. Progressive HER2 positive solid tumours (immunohistochemistry [IHC] positive or equivocal) with no available standard or curative treatment.
2. Eastern Cooperative Oncology Group (ECOG) performance score of 0-2.

Exclusion Criteria:

1. Active infectious disease considered by the Investigator to be incompatible with the protocol.
2. Patients not recovered from any therapy-related toxicities from previous therapies to at least CTCAE ≤ Grade 1 except in case of liver metastases or Gilbert's Syndrome or alopecia.
3. Brain metastases that are symptomatic or untreated or that require current therapy.
4. Previous treatment with immunotherapy within 8 weeks of starting study medication, chemotherapy, radiotherapy, molecular-targeted therapy, or biological therapies (including HER2 directed therapies) within 4 weeks of starting study medication, or hormone therapy within 2 weeks of starting study medication.
5. Use of any investigational drug within the past 4 weeks before start of study medication or concomitantly with this study except for investigational immune-stimulatory therapy (e.g. checkpoint-regulator targeted treatment). The minimum washout period should be 8 weeks before starting the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Maximal Tolerated Dose (MTD) of GBR 1302 | 28 Days
  Number of DLTs (dose limiting toxicities) after the first two administrations of study drug (i.e. Cycle 1) in each cohort
The relationship of the dose of GBR 1302 with the incidence, nature, and intensity of AEs according to CTCAEv4.03 | 28 Days

SECONDARY OUTCOMES:
Objective Response Rate (ORR) for solid tumors. | 2 cycles, 56 days
Disease control rate (DCR) for solid tumors | 2 cycles, 56 days
Duration of disease control (measured from drug start date to the date of disease progression or death for subjects who had CR or PR or SD during treatment). | At least 56 days
Maximum Concentration (Cmax) of GBR 1302 | 28 Days
Time to Maximum Concentration (Tmax) of GBR 1302 | 28 Days
Area Under Curve [AUC0-t and AUC0-tau] of GBR 1302 | 28 Days
Immunogenicity of GBR 1302 in terms of ADA formation assessed compared to baseline | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Khazan, MD, Study Director — Ichnos Sciences SA
Locations (8):
- United States (4):
  - Glenmark Investigational Site 204, Fairway, Kansas
  - Glenmark Investigational Site 209, Detroit, Michigan
  - Glenmark Investigational Site 201, Dallas, Texas
  - Glenmark Investigational Site 203, Salt Lake City, Utah
- Germany (4):
  - Glenmark Investigational Site 103, Berlin
  - Glenmark Investigational Site 102, Cologne
  - Glenmark Investigational Site 101, Dresden
  - Glenmark Investigational Site 104, Mainz